CLINICAL TRIAL: NCT01222572
Title: Stereotactic Boost for Locally Advanced Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual due to restrictive eligibility criteria
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Raymond H. Mak, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-240
Record Dates: First submitted 2010-10-08; First posted 2010-10-18 (Estimated); Results first posted 2014-09-05 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-05

CONDITIONS: Non-small Cell Lung Cancer; Lung Cancer; NSCLC
Keywords: radiation therapy; stereotactic radiotherapy; stereotactic boost
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Radiosurgery; Etoposide; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Stereotactic Boost to Chemoradiotherapy (Dose Level 1) (Experimental): Chemotherapy: Etoposide 50 mg/m2, d1-5, 29-33 and Cisplatin 50 mg/m2, d1, 8, 29, 36; Conventional RT Dose to Primary: 54 Gy; Stereotactic Boost to Primary: 10 Gy; Total Dose to Primary: 64 Gy
  - Patients were to start radiation to the primary tumor site and to the lymph nodes and chemotherapy in the same week. The treatment was identical to standard chemotherapy and radiation treatment until the 5th week. During the fifth week, patents would undergo another radiation mapping session to prepare for the stereotactic boost. After that, the radiation treatments to the lymph nodes would continue but the radiation treatment to the primary cancer site would stop until the last week (week 7). During week 7, participants would receive 2 doses of stereotactic radiotherapy to the site of the primary tumor instead of the lower doses of radiotherapy that they were treated with up to that point.
  Interventions: Radiation: Stereotactic boost; Radiation: Conventional RT; Drug: Etoposide; Drug: Cisplatin
- Stereotactic Boost to Chemoradiotherapy (Dose Level 2) (Experimental): Chemotherapy: Etoposide 50 mg/m2, d1-5, 29-33 and Cisplatin 50 mg/m2, d1, 8, 29, 36; Conventional RT Dose to Primary: 50 Gy; Stereotactic Boost to Primary: 15 Gy; Total Dose to Primary: 65 Gy
  - Patients were to start radiation to the primary tumor site and to the lymph nodes and chemotherapy in the same week. The treatment was identical to standard chemotherapy and radiation treatment until the 5th week. During the fifth week, patents would undergo another radiation mapping session to prepare for the stereotactic boost. After that, the radiation treatments to the lymph nodes would continue but the radiation treatment to the primary cancer site would stop until the last week (week 7). During week 7, participants would receive 2 doses of stereotactic radiotherapy to the site of the primary tumor instead of the lower doses of radiotherapy that they were treated with up to that point.
  Interventions: Radiation: Stereotactic boost; Radiation: Conventional RT; Drug: Etoposide; Drug: Cisplatin
- Stereotactic Boost to Chemoradiotherapy (Dose Level 3) (Experimental): Chemotherapy: Etoposide 50 mg/m2, d1-5, 29-33 and Cisplatin 50 mg/m2, d1, 8, 29, 36; Conventional RT Dose to Primary: 46 Gy; Stereotactic Boost to Primary: 20 Gy; Total Dose to Primary: 66 Gy
  - Patients were to start radiation to the primary tumor site and to the lymph nodes and chemotherapy in the same week. The treatment was identical to standard chemotherapy and radiation treatment until the 5th week. During the fifth week, patents would undergo another radiation mapping session to prepare for the stereotactic boost. After that, the radiation treatments to the lymph nodes would continue but the radiation treatment to the primary cancer site would stop until the last week (week 7). During week 7, participants would receive 2 doses of stereotactic radiotherapy to the site of the primary tumor instead of the lower doses of radiotherapy that they were treated with up to that point.
  Interventions: Radiation: Stereotactic boost; Radiation: Conventional RT; Drug: Etoposide; Drug: Cisplatin

INTERVENTIONS:
Radiation: Stereotactic boost
  Other Names: Stereotactic Body Radiotherapy (SBRT)
Radiation: Conventional RT
Drug: Etoposide
Drug: Cisplatin

SUMMARY:
In this research study the investigators are looking for the highest dose of a stereotactic radiation boost that can be given safely. Because stereotactic radiation is so precise, the investigators are testing whether it can be used to increase the dose to the primary tumor without significantly increasing the side effects the participant experiences; the goal is to improve the likelihood of killing the tumor.

DETAILED DESCRIPTION:
Primary Objectives Phase I: Determination of the MTD and dose-limiting toxicities of a stereotactic boost to chemoradiotherapy for stage II/III non-small cell lung cancer.

Phase II: Two-year local control rate

Secondary Objectives

* To evaluate the safety and tolerability of a stereotactic boost to chemoradiotherapy.
* To determine the 2-year overall survival.
* To determine the 2-year disease-free survival.
* To determine the 2-year regional control rate.
* To characterize the change in pulmonary function tests over the first 2 years after chemoradiotherapy.

Statistical Design The Phase I study followed a standard 3+3 dose escalation design. Three dose levels were evaluated. The DLT observation period was the 7-week chemoradiotherapy period and the subsequent 8-week recovery period.

To better study the toxicity at the MTD of the stereotactic boost, there was a 10 patient expansion cohort.The primary endpoint of the phase II portion of the study was two-year local failure rate of the protocol treatment. Local failure was defined as biopsy-proven recurrent disease, or if a biopsy was not attainable, by increasing FDG-avidity on PET-CT on 2 consecutive scans at least 1 month apart. Based on prior studies, a 2-year local failure rate of 15% would be worthy of further study, while a 2-year local failure rate of 35% would not justify further utilization of the treatment. With 32 eligible patients on this study, the treatment will be deemed promising if at least 25 patients are free of local failure at 2 years. Using this design, there was an 8% probability of declaring the treatment worthy of further study if the true 2-year local failure rate was 35%, and a 90% probability of declaring the treatment worthy of further study if the true 2-year local failure rate was 15% by using a one-sided one-sample exact binomial test.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage II or stage III non-small cell lung cancer, or stage IV non-small cell lung cancer that will be treated with curative intent
* Evaluated by a surgeon and deemed inoperable
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension as 10mm or greater with chest CT scan.
* No active malignancy within the past 5 years, except for non-melanoma skin cancers or carcinoma in situ of the cervix
* 18 years or older
* Life expectancy of greater then 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Normal organ and marrow function as outlined in the protocol
* Forced expiratory volume (FEV1) of 1 L or greater OR 50% or greater of predicted

Exclusion Criteria:

* Primary tumor size greater then 6cm
* Prior history of thoracic radiotherapy
* May not be receiving any other study agents
* History of pulmonary fibrosis
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cisplatin or etoposide
* Primary tumor < 1.5 cm beyond hilar lymphadenopathy (if any) and 1.5 cm from proximal bronchial tree, defined as the trachea, right and left mainstem bronchus, and lobar bronchi until the 1st lobar segment
* Uncontrolled intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breast feeding women
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin
* Human immunodeficiency virus (HIV)-positive individuals on combination antiretroviral therapy
* Patients who are planned to receive the following medication: granulocyte colony-stimulating factor (G-CSF), bevacizumab, cetuximab, cyclosporine, anti-tumor necrosis factor agents, amifostine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-12; Primary Completion 2012-03 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond H. Mak, MD, Principal Investigator — Dana-Farber Cancer Institute/Brigham and Women's Hospital
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to restrictive eligibility criteria, accrual did not meet expectations.
Groups:
- Stereotactic Boost to Chemoradiotherapy (Dose Level 1): Chemotherapy: Etoposide 50 mg/m2, d1-5, 29-33 and Cisplatin 50 mg/m2, d1, 8, 29, 36; Conventional RT Dose to Primary: 54 Gy; Stereotactic Boost to Primary: 10 Gy; Total Dose to Primary: 64 Gy
  Patients were to start radiation to the primary tumor site and to the lymph nodes and chemotherapy in the same week. The treatment was identical to standard chemotherapy and radiation treatment until the 5th week. During the fifth week, patents would undergo another radiation mapping session to prepare for the stereotactic boost. After that, the radiation treatments to the lymph nodes would continue but the radiation treatment to the primary cancer site would stop until the last week (week 7). During week 7, participants would receive 2 doses of stereotactic radiotherapy to the site of the primary tumor instead of the lower doses of radiotherapy that they were treated with up to that point.
- Stereotactic Boost to Chemoradiotherapy (Dose Level 2): Chemotherapy: Etoposide 50 mg/m2, d1-5, 29-33 and Cisplatin 50 mg/m2, d1, 8, 29, 36; Conventional RT Dose to Primary: 50 Gy; Stereotactic Boost to Primary: 15 Gy; Total Dose to Primary: 65 Gy
  Patients were to start radiation to the primary tumor site and to the lymph nodes and chemotherapy in the same week. The treatment was identical to standard chemotherapy and radiation treatment until the 5th week. During the fifth week, patents would undergo another radiation mapping session to prepare for the stereotactic boost. After that, the radiation treatments to the lymph nodes would continue but the radiation treatment to the primary cancer site would stop until the last week (week 7). During week 7, participants would receive 2 doses of stereotactic radiotherapy to the site of the primary tumor instead of the lower doses of radiotherapy that they were treated with up to that point.
- Stereotactic Boost to Chemoradiotherapy (Dose Level 3): Chemotherapy: Etoposide 50 mg/m2, d1-5, 29-33 and Cisplatin 50 mg/m2, d1, 8, 29, 36; Conventional RT Dose to Primary: 46 Gy; Stereotactic Boost to Primary: 20 Gy; Total Dose to Primary: 66 Gy
  Patients were to start radiation to the primary tumor site and to the lymph nodes and chemotherapy in the same week. The treatment was identical to standard chemotherapy and radiation treatment until the 5th week. During the fifth week, patents would undergo another radiation mapping session to prepare for the stereotactic boost. After that, the radiation treatments to the lymph nodes would continue but the radiation treatment to the primary cancer site would stop until the last week (week 7). During week 7, participants would receive 2 doses of stereotactic radiotherapy to the site of the primary tumor instead of the lower doses of radiotherapy that they were treated with up to that point.
Period: Overall Study
Arm/Group | Stereotactic Boost to Chemoradiotherapy (Dose Level 1) | Stereotactic Boost to Chemoradiotherapy (Dose Level 2) | Stereotactic Boost to Chemoradiotherapy (Dose Level 3)
Started | 1 | 0 | 0
Completed | 1 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Stereotactic Boost to Chemoradiotherapy (Dose Level 1)
Number analyzed (Participants) | 1
Age, Continuous [Mean (Full Range); unit: years] | 68 [68 to 68]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD is determined by the number of patients who experience a dose limiting toxicity (DLT). The MTD is defined as the highest dose at which fewer than one-third of patients experience a DLT. If no DLTs are observed, the MTD is not reached.
  DLTs were defined as follows (CTCAE v4.0):
  Grade 2 non-hematologic toxicities: Myelitis; Esophageal fistula, perforation, hemorrhage
  Grade 3 non-hematologic toxicities considered to be a direct result of therapy:
  Radiation pneumonitis; Pericarditis, pericardial effusion, pericardial tamponade; Esophageal necrosis, stenosis, ulcer; Dyspnea; Myelitis Grade 4 non-hematologic toxicities: Radiation pneumonitis; Pericarditis, pericardial effusion, pericardial tamponade; Esophagitis (not due to mediastinal irradiation unrelated to the stereotactic boost), esophageal necrosis, stenosis, ulcer; Dyspnea; Myelitis Grade 5 non-hematologic toxicity: Any
Time Frame: 7-week chemoradiotherapy period and the subsequent 8-week recovery period
Population: All treated participants who received at least one dose of the study drug and were evaluable for DLT.
Measure: Number; unit: participants with DLT
Arm/Group | Stereotactic Boost to Chemoradiotherapy (Dose Level 1)
Number analyzed (Participants) | 1
participants with DLT | 0

ADVERSE EVENTS:
Time Frame: Assessed from time of first dose, weekly during treatment, and through day 30 post treatment.
Arm/Group | Stereotactic Boost to Chemoradiotherapy (Dose Level 1)
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Study was closed due to poor accrual after enrollment of 1 patient and results of trial are not interpretable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No